CLINICAL TRIAL: NCT03936725
Title: Evaluation of Return to Work One Year After a Short Rehabilitation Program for Chronic Non Specific Low Back Pain Patients
Brief Title: Evaluation of Return to Work One Year After a Rehabilitation Program for Chronic Back Pain
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0166
Record Dates: First submitted 2019-04-26; First posted 2019-05-03 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Non Specific Chronic Low Back Pain
Keywords: Rehabilitation program; Non specific chronic low back pain; Return to work

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic and non specific low back pain patients: Chronic and non specific low back pain patients
  Interventions: Other: 1 year phone call : data collection

INTERVENTIONS:
Other: 1 year phone call : data collection — Included patients are contacted by telephone at 12 months after discharge. The investigators explain to the patient that this call is in the same context as a regular follow-up rehabilitation consultation and that the data collected will also be part of a study to evaluate and improve the program in which they participated. The interview will be transcribed in writing in their computerized and secure medical file. During this 20-minute telephone conversation, the patient answers a number of questions via a standardized questionnaire, in order to gather the various criteria for judgment.
  If patients do not answer the first call, a phone message will be left and they will be contacted again up to 2 times. Patients who do not respond to 3 calls will be considered lost to follow-up.

SUMMARY:
Return to work is one of the essential objectives of functional spinal restoration programs. When the duration of the work stoppage increases, the chances of returning to work become worse. No studies have yet evaluated the value of a short 2-week restoration program.

The purpose of this study is to determine whether a 2-week functional restoration program regains a return-to-work rate similar to longer-term restoration programs at one year post-program.

This retrospective study with prospective referral included 200 patients with non specific chronic low-back pain who participated in a self-care rehabilitation program between May 2018 and May 2019. The program included both physical and educational approaches to dealing with the condition. The duration was two weeks with follow-up at three months.

The main evaluation criterion was to evaluate the return to work rate by telephone at one year post-program. Secondary objectives were to observe return-to-work conditions, absenteeism, recovery time, pain and physical activity at one year post-program and also to observe if there was a possible association between intrinsic/extrinsic factors and return to work

DETAILED DESCRIPTION:
Patients were included in the study from May 2019 to May 2020 if they had chronic nonspecific low back pain of more than 12 weeks according to the French health authority (High Authority of Health).

The data for this study were collected after validation by the ethics committee (Institutional Review Board). Initial data were collected from generation of a list of computerized medical records of low back pain patients who participated in the program between May 2018 and May 2019 and were hospitalized in the day or week area of follow-up and rehabilitative care : age, sex, BMI, marital status, clinical elements related to the low-back pain (total duration of low back pain, history of spine surgery, last spinal imaging, pain measured on a visual analog scale, analgesic consumption, tobacco consumption, physical activity, self-exercise, physiotherapy, Schober index, finger-ground distance, poplitates angles, heel-buttock distance) and professional situation (professional status, carrying heavy loads, sick leave accumulated prior hospitalization for back pain, professional status, occupational disease, occupational accident, disability, half-time therapy).

One-year post-program data were collected by telephone after consent was received. The investigators collected the date of return to work, elements concerning the conditions of return to work (modification of the previous position, working time, type of contract, work stoppages related to back pain, evolution of global job satisfaction before/after program ) and clinical elements (change in pain after the program, physical activity, self-stretching exercises, spine operation after the program,satisfaction of the rehabilitation program, benefit provided by the program).

Reference Methodology MR-004 was applied to the study after approval by the Data Protection Officer (CNIL). An information letter was sent to the selected patients to comply with the applicable regulations (RGPD). The patient was not included if he returned the non-consent form.

Program : The duration of hospitalization was 2 weeks and the care program was delivered, for each patient, by the same medical and paramedical team including doctors, physiotherapists, occupational therapists, a nurse. There was no change in the program during the 2018-2019 year, so the hospitalized patients received the same program. The functional restoration program included stretching and muscle strengthening of the spine and sub-pelvic planes, abdominal sheathing, gymnastics, exercise re-training sessions, self-exercise training, balneotherapy, relaxation sessions, sessions of body awareness and ergonomics.

ELIGIBILITY:
Inclusion criteria

* age between 18 and 65 years
* lumbalgia for more than 12 weeks labeled nonspecific (= common mechanics)
* have benefited fully from the 2-week day hospital rehabilitation program.

Exclusion criteria

* secondary low back pain
* immediate postoperative hospitalization (<3 months)
* patient who died at the time of the study
* non-updated telephone numbers
* housewife, students subject subject to protection (curatorship, safeguard of justice, guardianship)
* Serious co-morbidities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who participated in the functional spine rehabilitation program proposed by the department of Physical Medicine and Rehabilitation of the University Hospital of Lapeyronie in Montpellier
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Return to work at one year post-program | 1 year
  code yes/no in the questionnaire with date of return to work after program.

SECONDARY OUTCOMES:
Absenteeism rate during the 12-month post-program | 1 year
  Absenteeism rate during the 12-month post-program evaluated in days by the questionnaire with suggested answers
The delay of return to work post-program | 1 year
  The delay of return to work post-program evaluated in the day by the questionnaire with suggestion of answers
Conditions of return to work | 1 year
  Conditions of return to work evaluated by several items of the questionnaire with suggested answers
Pain at 1 year post-program | 1 year
  Pain at 1 year post-program evaluated by a numerical scale (EVA)
Physical activity at 1 year post-program | 1 year
  Physical activity at 1 year post-program evaluate by code yes / no
Evaluating intrinsic or extrinsic factors are associated with a professional recovery | 1 year
  evaluate whether certain intrinsic and / or extrinsic factors are possibly associated favorably with a professional recovery

CONTACTS AND LOCATIONS:
Overall Officials: Marie HILLION, medical intern, Principal Investigator — CHU de Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC